CLINICAL TRIAL: NCT06904729
Title: An Exploratory Clinical Study of the Safety and Efficacy of CAR-T in Children With Refractory/Recurrent Lupus Nephritis Disease
Brief Title: Chimeric Antigen Receptors T Cells for Refractory/Recurrent Lupus Nephritis in Children
Acronym: CAR-T
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2025]040A01
Record Dates: First submitted 2025-02-26; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-02

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental): Children who met the inclusion criteria were given transfusions of CAR-T cells
  Interventions: Biological: Low-dose CAR-T cells group; Biological: High-dose CAR-T cells group

INTERVENTIONS:
Biological: Low-dose CAR-T cells group — This group of patients received low dose novel structure of Chimeric Antigen Receptors T (CAR-T) cells therapy with an infusion dose of approximately 5×100,000 cells/Kg.
Biological: High-dose CAR-T cells group — This group of patients received high dose novel structure of Chimeric Antigen Receptors T (CAR-T) cells therapy with an infusion dose of approximately 1×1000,000 cells/Kg.

SUMMARY:
The goal of this prospective, open, single-arm clinical trial was to evaluate the safety and potential efficacy of CAR T cell therapy in children with refractory/recurrent lupus nephritis. The persistence and cell phenotype of CAR-T cells in vivo and CAR-T treatment-related inflammatory factors were evaluated after treatment. To explore new therapeutic methods, in order to reduce the side effects of traditional therapeutic drugs, increase curative effect, and finally make patients obtain long-term survival and improve survival quality.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-18 years old (including critical value);
2. Diagnosed with SLE according to the 2019 EULAR/ACR SLE classification criteria;
3. According to the 2018 ISN/RPS LN standards diagnosed with active Class III or IV LN, with or without a membranous component and the biopsy must be performed within 6 months prior to screening;
4. SLEDAI-2000 score ≥8 points;
5. Meeting the diagnosis of refractory lupus nephritis,

   1. defined as treatment with two or more immunosuppressants (including glucocorticoids, cyclophosphamide, tacrolimus, mycophenolic acid analogues, leflunomide, and cyclosporine) for more than 6 months without inducing remission or relapse after remission,
   2. accompanied by proteinuria without remission;
6. Positive expression of CD19 in peripheral blood B cells determined by flow cytometry;
7. Participants had good venous access, no contraindications for cell collection;
8. Participants and their guardians sign the informed consent, understand the study procedures and participate in the clinical study voluntarily;
9. The functions of important organs are basically normal:

   1. Hematopoietic function (blood routine should meet):

      * Lymphocyte count ≥1×109/L,
      * White blood cell count ≥3×109/L,
      * Neutrophil count ≥1×109/L (no colony-stimulating factor treatment within 2 weeks prior to examination),
      * Hemoglobin ≥60g/L;
   2. Liver function:

      * ALT≤3×ULN (except elevated ALT caused by inflammatory myopathy),
      * AST≤3×ULN (except for elevated AST caused by inflammatory myopathy),
      * TBIL≤1.5×ULN (except Gilbert syndrome, total bilirubin ≤3.0×ULN);
   3. Renal function: eGFR ≥30 ml/(min.1.73m2) (Schwartz formula, except abnormal renal function by SLE);
   4. Coagulation function:

      * International standardized ratio (INR) ≤1.5×ULN,
      * prothrombin time (PT) ≤1.5×ULN;
   5. Heart function: hemodynamic stability;
10. Anti-nuclear antibody (ANA) ≥1:80;
11. Eastern Cancer Cooperation Group (ECOG) physical status score 0 to 2.

Exclusion Criteria:

1. Received kidney transplant previously;
2. Serious drug allergy history or allergy;
3. Presence or suspicion of fungal, bacterial, viral or other infections that cannot be controlled or require treatment;
4. Complicated with severe organ dysfunction of heart, liver, lung or coagulation dysfunction;
5. Complicated with congenital immunoglobulin deficiency;
6. Participants with infectious diseases:

   1. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBc Ab) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range;
   2. Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range;
   3. Human immunodeficiency virus (HIV) antibody positive;
   4. Syphilis positive;
7. Diagnosed with malignant tumors in the last five years.
8. Suffer from severe central nervous system disease, mental illness and severe cognitive dysfunction;
9. Participated in other clinical trials within 3 months before enrollment;
10. Received CAR-T therapy previously;
11. Other situations that the researcher considers unsuitable for inclusion.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with CAR-T cells treatment-related adverse events(AE) | 2 years
  Incidence and severity of treatment-related AE, including adverse event of special interest (AESI), as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Overall renal response (ORR) rete | 2 years
  ORR rate: Number of participants meet the complete renal response (CRR) or partial renal response (PRR) as a percentage of total participants. Follow-up for 2 years after CAR-T cells reinfusion, monitored and recorded ORR at study set time points (Month 3, Month 6, Month 12, Month 24, or participant withdrawal from the study).
Number of participants with SRI-4 response | 2 years
  Number of participants with SLE response Index 4(SRI-4) response: including Systemic Lupus Erythematosus Disease Activity Index(SLEDAI) 2000 scores decreased by ≥4 points from baseline, PGA with no worsening (VAS increased by <0.30 points from baseline), British Isles Lupus Assessment Group(BILAG) 2004 with no new A domain score and no more than 1 new B domain scores. Follow-up for 2 years after CAR-T cells reinfusion, monitored and recorded SRI-4 response at study set time points (Month 3, Month 6, Month 12, Month 24, or participant withdrawal from the study).

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women and Children Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No